CLINICAL TRIAL: NCT01299389
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dose, Multicenter Study of JNS010 (Paliperidone Palmitate) in Patients With Schizophrenia
Brief Title: An Efficacy and Safety Study of Paliperidone Palmitate in Participants With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017026; PALM-JPN-4 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-01-27; First posted 2011-02-18 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Schizophrenia
Keywords: Paliperidone palmitate; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paliperidone palmitate (Experimental)
  Interventions: Drug: Paliperidone palmitate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paliperidone palmitate — Paliperidone palmitate will be given intramuscularly as an initial loading dose of 150 milligram (mg) equivalents (eq.) on Day 1 and 100 mg eq. on Day 8, followed by 75 mg eq. on Day 36 and Day 64. Participants who complete double-blind period or discontinued early from double-blind period will have follow-up visits during post-observational period at Weeks 4, 8 and 12 after the last injection in the double-blind period. Participants will not receive any study drug during post-observational period.
  Arms: Paliperidone palmitate
Drug: Placebo — Matching Placebo will be given intramuscularly (Injection of a drug into a muscle) on Day 1, Day 8, Day 36 and Day 64. Participants who complete double-blind period or discontinued early from double-blind period will have follow-up visits during post-observational period at Weeks 4, 8 and 12 after the last injection in the double-blind period. Participants will not receive any study drug during post-observational period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of paliperidone palmitate as compared with placebo in the treatment of participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions [a false belief held in the face of strong differing evidence, especially as a symptom of psychiatric disorder] and hallucinations [imagining things], and withdrawal into the self).

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), double-blind (neither physician nor participant knows the name of the assigned drug), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect), parallel-group (comparing the response in two groups of participants receiving different treatments), fixed-dose, multi-center (when more than one hospital or medical school team work on a medical research study) study of paliperidone palmitate in participants with schizophrenia. The study will consist of 3 periods: an up to 2-week pre-observation (screening) period, a double-blind period from Day 1 (baseline) to Week 13 (end of double-blind period) assessment, and a post-observation period starting after the Week 13 assessment to Week 21. For participants who discontinue the study before the last assessment in Week 13, the post-observation period will start after the discontinuation from double-blind period assessment with follow-up visits at 4, 8, and 12 weeks after the last injection. After completion of the double-blind period (Week 13), discontinuation of double-blind period treatment or withdrawal from the study, participants may receive treatment consistent with the usual standard of care. The total duration of the study will be 21 weeks, including the double-blind and post-observation periods. Participants will be randomly assigned to 1 of 2 treatment groups in a 1:1 ratio (intramuscular injections of either paliperidone palmitate or matching placebo). Injections of paliperidone palmitate or placebo will be given at Day 1 and at Weeks 1, 5, and 9 by a study drug manager and/or injector. For those participants receiving paliperidone palmitate, the Day 1 injection will be 150 milligram equivalent (mg eq.) paliperidone palmitate, followed by 100 mg eq. injections of paliperidone palmitate at Week 1, and 75 mg eq. injections of paliperidone palmitate at Weeks 5 and 9. Participants randomly assigned to placebo will receive injections matching the paliperidone palmitate injections on the same days. Efficacy will be assessed using Positive and Negative Syndrome Scale (PANSS), Clinical Global Impression - Severity (CGI-S). Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants meeting Diagnostic criteria for schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision
* Women had to be: postmenopausal (for at least 2 years), surgically sterile (had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), abstinent (as judged by the investigator; per local regulations), or if sexually active, be practicing a highly effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [eg, condoms, diaphragm, or cervical cap, with spermicidal foam, cream, or gel], male partner sterilization) as local regulations permitted, before entry, and had to agree to continue to use the same method of contraception throughout the study
* A Positive and Negative Syndrome Scale (PANSS) total score at screening and at baseline (Day 1) of 60 to 120
* Documented history of exposure to either a risperidone formulation or a paliperidone formulation and known to be tolerated before baseline (Day 1) (Even if the participant's experience of taking risperidone or paliperidone cannot be confirmed at the time of informed consent, the participant will be able to meet this criterion if the participant takes oral risperidone 2 mg/day or more or paliperidone ER 6 mg/day or more for at least 4 days between the day of informed consent and the day before baseline, and it is possible to confirm that there is no lack of tolerability in the participant)
* Women of childbearing potential must have a negative beta human chorionic gonadotropin pregnancy test at the screening urine pregnancy test

Exclusion Criteria:

* Primary active Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision Axis I diagnosis other than schizophrenia
* A Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision diagnosis of active substance dependence within 3 months before screening (nicotine and caffeine are not exclusionary)
* Relevant history or current presence of any significant or unstable cardiovascular, respiratory, neurological (including seizures or significant cerebrovascular), renal, hepatic, hematologic, endocrine, immunologic, or other systemic disease
* History or current presence of neuroleptic malignant syndrome or tardive dyskinesia
* Known or suspected hypersensitivity or intolerance to risperidone, paliperidone, Intralipid, or any of their excipients (including egg yolks, soybean oil, phospholipids, and glycerol)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (56):
- Japan (40):
  - Fujioka
  - Fujisawa
  - Fukui
  - Fukuoka
  - Hadano
  - Ichikawa
  - Itoman
  - Kanzaki
  - Kashihara
  - Kasuya
  - Kawasaki
  - Kitagunma
  - Kitakyushu
  - Kobe
  - Kodaira
  - Koshigaya
  - Kumagaya
  - Kumamoto
  - Kurayoshi
  - Kure
  - Kurume
  - Mitaka
  - Miyazaki
  - Moriguchi
  - Nanyō
  - Nishinomiya
  - Ohta
  - Okinawa
  - Oyabe
  - Sakai
  - Shibukawa
  - Takatsuki
  - Tamana
  - Tokyo
  - Toyama
  - Toyoake
  - Urasoe
  - Yatsushiro
  - Yokkaichi
  - Yokohama
- South Korea (9):
  - Busan
  - Chungcheongbuk-Do
  - Daegu
  - Deajun
  - Incheon
  - Inchun
  - Jeonju
  - Seongnam
  - Seoul
- Taiwan (7):
  - Bali Township, Taipei County
  - Changhua
  - Hualien City
  - Kaohsiung City
  - Tainan
  - Taipei
  - Taoyuan District

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Double-blind): Matching Placebo was given intramuscularly (Injection of a drug into a muscle) on Day 1, Day 8, Day 36 and Day 64.
- Paliperidone Palmitate (Double-blind): Paliperidone palmitate was given intramuscularly as an initial loading dose of 150 milligram (mg) equivalents (eq.) on Day 1 and 100 mg eq. on Day 8, followed by 75 mg eq. on Day 36 and Day 64.
- Placebo (Post-observational); Paliperidone Palmitate (Post-observational): Participants who completed double-blind period or discontinued early from double-blind period had follow-up visits during post-observational period at Weeks 4, 8 and 12 after the last injection in the double-blind period. Participants did not receive any study drug during post-observational period.
Period: Double-blind
Arm/Group | Placebo (Double-blind) | Paliperidone Palmitate (Double-blind) | Placebo (Post-observational) | Paliperidone Palmitate (Post-observational)
Started | 164 | 159 | 0 | 0
Completed | 55 | 95 | 0 | 0
Not Completed | 109 | 64 | 0 | 0
Not completed — Adverse Event | 45 | 27 | 0 | 0
Not completed — Lack of Efficacy | 45 | 21 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 13 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0
Not completed — fail to meet "study population" criteria | 0 | 1 | 0 | 0
Period: Post-observational
Arm/Group | Placebo (Double-blind) | Paliperidone Palmitate (Double-blind) | Placebo (Post-observational) | Paliperidone Palmitate (Post-observational)
Started | 0 | 0 | 156 | 155
Completed | 0 | 0 | 144 | 149
Not Completed | 0 | 0 | 12 | 6
Not completed — Other | 0 | 0 | 12 | 6

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomly assigned participants who received at least 1 injection of double-blind study drug.
Groups:
- Placebo (Double-blind): Matching Placebo was given intramuscularly (Injection of a drug into a muscle) on Day 1, Day 8, Day 36 and Day 64. Participants who completed double-blind period or discontinued early from double-blind period had follow-up visits during post-observational period at Weeks 4, 8 and 12 after the last injection in the double-blind period. Participants did not receive any study drug during post-observational period.
- Paliperidone Palmitate (Double-blind): Paliperidone palmitate was given intramuscularly as an initial loading dose of 150 milligram (mg) equivalents (eq.) on Day 1 and 100 mg eq. on Day 8, followed by 75 mg eq. on Day 36 and Day 64. Participants who completed double-blind period or discontinued early from double-blind period had follow-up visits during post-observational period at Weeks 4, 8 and 12 after the last injection in the double-blind period. Participants did not receive any study drug during post-observational period.
- Total: Total of all reporting groups
Arm/Group | Placebo (Double-blind) | Paliperidone Palmitate (Double-blind) | Total
Number analyzed (Participants) | 164 | 159 | 323
Age Continuous [Mean (Standard Deviation); unit: years] | 44.0 (12.41) | 45.7 (13.55) | 44.8 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 58 | 139
  Male | 83 | 101 | 184

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score at Week 13 or Early Discontinuation
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210, higher scores indicate worsening.
Time Frame: Baseline and Week 13 or early discontinuation
Population: Full Analysis Set (FAS) population included all randomly assigned participants who received at least 1 injection of double-blind study drug and had baseline and at least 1 post-baseline PANSS total scores. Last Observation Carried Forward (LOCF) method was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo (Double-blind): Matching Placebo was given intramuscularl (Injection of a drug into a muscle) on Day 1, Day 8, Day 36 and Day 64.
Arm/Group | Placebo (Double-blind) | Paliperidone Palmitate (Double-blind)
Number analyzed (Participants) | 164 | 158
units on a scale
  Baseline | 83.5 (15.18) | 85.7 (14.57)
  Change at Week 13 or Early Discontinuation | 6.9 (19.13) | -3.1 (20.32)
Statistical Analysis 1: Comparison: Placebo (Double-blind) vs Paliperidone Palmitate (Double-blind); Change at Week 13 or Early Discontinuation: P value were calculated using an analysis of covariance (ANCOVA) model with treatment and country as factors and baseline PANSS total score as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least squares (LS) means difference = -9.7, 95% CI 2-sided [-14.0 to -5.4], Standard Error of Mean 2.19

2. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Week 13 or Early Discontinuation
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants", higher scores indicate worsening.
Time Frame: Baseline and Week 13 or early discontinuation
Population: FAS population included all randomly assigned participants who received at least 1 injection of double-blind study drug and had baseline and at least 1 post-baseline PANSS total scores. LOCF method was used.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Placebo (Double-blind): Matching Placebo was given intramuscularly on Day 1, Day 8, Day 36 and Day 64.
Arm/Group | Placebo (Double-blind) | Paliperidone Palmitate (Double-blind)
Number analyzed (Participants) | 164 | 158
units on a scale
  Baseline | 4.0 [2 to 7] | 4.0 [2 to 6]
  Change at Week 13 or Early Discontinuation | 0.0 [-3 to 3] | 0.0 [-3 to 3]

3. Secondary Outcome: Participants With Response to the Treatment as Per PANSS Total Score.
Description: Participants with response were defined as those participants who shows 30 percent or more and 20 percent or more reduction in PANSS total score.
Time Frame: up to Week 13 or early discontinuation
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo (Double-blind) | Paliperidone Palmitate (Double-blind)
Number analyzed (Participants) | 164 | 158
participants
  Greater than or equal to 30 percent Improvement | 14 | 36
  Greater than or equal to 20 percent Improvement | 23 | 52

4. Secondary Outcome: Change From Baseline in PANSS Marder Subscale Scores at Week 13 or Early Discontinuation
Description: The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). Positive symptoms subscale consists of 8 items with total score range of 8-56; negative symptoms subscale and disorganized thoughts subscale, each consists of 7 items with total score range of 7-49, uncontrolled hostility/excitement subscale and anxiety/depression subscale, each consists of 4 items with total score range of 4-28, higher score indicates greater severity.
Time Frame: Baseline and Week 13 or early discontinuation (ED)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind) | Paliperidone Palmitate (Double-blind)
Number analyzed (Participants) | 164 | 158
units on a scale
  Positive symptoms: Baseline | 24.3 (5.56) | 24.2 (5.66)
  Positive symptoms: Change at Week 13 or ED | 1.6 (6.06) | -1.1 (6.29)
  Negative symptoms: Baseline | 21.7 (6.22) | 22.8 (6.04)
  Negative symptoms: Change at Week 13 or ED | 0.9 (5.82) | -1.4 (5.76)
  Disorganized thoughts: Baseline | 19.6 (5.13) | 20.8 (4.83)
  Disorganized thoughts: Change at Week 13 or ED | 1.9 (5.24) | -0.6 (5.11)
  Uncontrolled hostility/excitement: Baseline | 8.3 (3.07) | 8.6 (3.42)
  Uncontrolled hostility: Change at Week 13 or ED | 1.9 (4.23) | 0.4 (4.15)
  Anxiety/depression: Baseline | 9.5 (3.02) | 9.4 (3.14)
  Anxiety/depression: Change at Week 13 or ED | 0.7 (3.27) | -0.4 (3.54)
Statistical Analysis 1: Comparison: Placebo (Double-blind) vs Paliperidone Palmitate (Double-blind); Positive symptoms (change at Week 13 or ED): P value was calculated using an ANCOVA model with treatment and country as factors and baseline PANSS factor scores as covariates; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean difference = -2.7, 95% CI 2-sided [-4.1 to -1.4], Standard Error of Mean 0.69
Statistical Analysis 2: Comparison: Placebo (Double-blind) vs Paliperidone Palmitate (Double-blind); Negative symptoms (change at Week 13 or ED): P value was calculated using an ANCOVA model with treatment and country as factors and baseline PANSS factor scores as covariates; Test type: Superiority or Other; p = 0.0012, ANCOVA; LS Mean difference = -2.0, 95% CI 2-sided [-3.2 to -0.8], Standard Error of Mean 0.61
Statistical Analysis 3: Comparison: Placebo (Double-blind) vs Paliperidone Palmitate (Double-blind); Disorganized thoughts (change at Week 13 or ED): P value was calculated using an ANCOVA model with treatment and country as factors and baseline PANSS factor scores as covariates; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean difference = -2.2, 95% CI 2-sided [-3.4 to -1.1], Standard Error of Mean 0.57
Statistical Analysis 4: Comparison: Placebo (Double-blind) vs Paliperidone Palmitate (Double-blind); Uncontrolled hostility/excitement (change at Week 13 or ED): P value was calculated using an ANCOVA model with treatment and country as factors and baseline PANSS factor scores as covariates; Test type: Superiority or Other; p = 0.0023, ANCOVA; LS Mean difference = -1.4, 95% CI 2-sided [-2.3 to -0.5], Standard Error of Mean 0.45
Statistical Analysis 5: Comparison: Placebo (Double-blind) vs Paliperidone Palmitate (Double-blind); Anxiety/depression (change at Week 13 or ED): P value was calculated using an ANCOVA model with treatment and country as factors and baseline PANSS factor scores as covariates; Test type: Superiority or Other; p = 0.0025, ANCOVA; LS Mean difference = -1.1, 95% CI 2-sided [-1.9 to -0.4], Standard Error of Mean 0.37

5. Secondary Outcome: Change From Baseline in PANSS Negative Subscale Score at Week 13 or Early Discontinuation
Description: Negative Syndrome Scale (range 7-49): Sum of scores for items 1-7 in negative subscale: blunted effect, emotional withdrawal, poor rapport, passive apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking, higher scores indicate worsening.
Time Frame: Baseline and Week 13 or early discontinuation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind) | Paliperidone Palmitate (Double-blind)
Number analyzed (Participants) | 164 | 158
units on a scale
  Baseline | 22.7 (6.19) | 24.0 (5.77)
  Change at Week 13 or Early Discontinuation | 0.9 (5.54) | -1.5 (5.38)
Statistical Analysis 1: Comparison: Placebo (Double-blind) vs Paliperidone Palmitate (Double-blind); Change at Week 13 or Early Discontinuation: P value were calculated using an ANCOVA model with treatment and country as factors and baseline PANSS total score as a covariate; Test type: Superiority or Other; p = 0.0003, ANCOVA; LS Mean difference = -2.1, 95% CI 2-sided [-3.3 to -1.0], Standard Error of Mean 0.59

6. Secondary Outcome: Change From Baseline in PANSS Positive Subscale Score at Week 13 or Early Discontinuation
Description: Positive Syndrome Scale (range 7-49): Sum of scores for items 1-7 in positive subscale: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility, higher scores indicate worsening.
Time Frame: Baseline and Week 13 or early discontinuation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind) | Paliperidone Palmitate (Double-blind)
Number analyzed (Participants) | 164 | 158
units on a scale
  Baseline | 19.3 (4.97) | 19.5 (5.47)
  Change at Week 13 or Early Discontinuation | 2.2 (5.82) | -0.6 (6.19)
Statistical Analysis 1: Comparison: Placebo (Double-blind) vs Paliperidone Palmitate (Double-blind); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean difference = -2.8, 95% CI 2-sided [-4.1 to -1.5], Standard Error of Mean 0.67

7. Secondary Outcome: Change From Baseline in PANSS General Psychopathology Subscale Score at Week 13 or Early Discontinuation
Description: General Psychopathology (range 16-112): Sum of scores for somatic concern, anxiety, guilt feelings, tension, mannerisms/posturing, depression, motor retardation, uncooperativeness, unusual thought content, disoriented, poor attention, lack of judgment/insight, disturbance of volition, poor impulse control, preoccupation, and active social avoidance, higher scores indicate worsening.
Time Frame: Baseline and Week 13 or early discontinuation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind) | Paliperidone Palmitate (Double-blind)
Number analyzed (Participants) | 164 | 158
units on a scale
  Baseline | 41.4 (7.97) | 42.3 (7.85)
  Change at Week 13 or Early Discontinuation | 3.8 (10.32) | -1.0 (11.04)
Statistical Analysis 1: Comparison: Placebo (Double-blind) vs Paliperidone Palmitate (Double-blind); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean difference = -4.6, 95% CI 2-sided [-6.9 to -2.3], Standard Error of Mean 1.17

ADVERSE EVENTS:
Time Frame: From signing of the informed consent until study completion.
Groups:
- Paliperidone Palmitate (Post-0bservational): Participants who completed double-blind period or discontinued early from double-blind period had follow-up visits during post-observational period at Weeks 4, 8 and 12 after the last injection in the double-blind period. Participants did not receive any study drug during post-observational period.
Arm/Group | Placebo (Double-blind) | Paliperidone Palmitate (Double-blind) | Placebo (Post-observational) | Paliperidone Palmitate (Post-0bservational)
Serious Adverse Events (participants affected / at risk) | 25/164 | 10/159 | 4/156 | 6/155
Other Adverse Events (participants affected / at risk) | 131/164 | 133/159 | 94/156 | 79/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind) (N=164) | Paliperidone Palmitate (Double-blind) (N=159) | Placebo (Post-observational) (N=156) | Paliperidone Palmitate (Post-0bservational) (N=155)
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Psychiatric symptom (Psychiatric disorders) | 13 | 4 | 2 | 2
Schizophrenia (Psychiatric disorders) | 3 | 4 | 2 | 2
Suicide attempt (Psychiatric disorders) | 2 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Self injurious behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind) (N=164) | Paliperidone Palmitate (Double-blind) (N=159) | Placebo (Post-observational) (N=156) | Paliperidone Palmitate (Post-0bservational) (N=155)
Nasopharyngitis (Infections and infestations) | 10 | 20 | 13 | 13
Upper respiratory tract infection (Infections and infestations) | 7 | 8 | 4 | 6
Cystitis (Infections and infestations) | 0 | 2 | 0 | 1
Hordeolum (Infections and infestations) | 2 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 3 | 1
Adenoviral conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 5 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Diet refusal (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperphagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 25 | 27 | 6 | 6
Psychiatric symptom (Psychiatric disorders) | 33 | 14 | 4 | 2
Anxiety (Psychiatric disorders) | 13 | 10 | 5 | 1
Aggression (Psychiatric disorders) | 1 | 4 | 0 | 1
Agitation (Psychiatric disorders) | 4 | 1 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 2 | 2 | 1 | 0
Delusion (Psychiatric disorders) | 1 | 2 | 0 | 1
Persecutory delusion (Psychiatric disorders) | 2 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 2 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 2 | 0 | 1 | 0
Self injurious behaviour (Psychiatric disorders) | 2 | 0 | 1 | 0
Anger (Psychiatric disorders) | 0 | 1 | 0 | 0
Catatonia (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 2
Emotional disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Hostility (Psychiatric disorders) | 0 | 1 | 0 | 0
Inappropriate affect (Psychiatric disorders) | 1 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Obsessive thoughts (Psychiatric disorders) | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Soliloquy (Psychiatric disorders) | 1 | 0 | 0 | 0
Somatic delusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Impulse-control disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 8 | 16 | 6 | 1
Headache (Nervous system disorders) | 6 | 8 | 5 | 4
Akathisia (Nervous system disorders) | 3 | 8 | 11 | 5
Dizziness (Nervous system disorders) | 5 | 1 | 4 | 1
Tremor (Nervous system disorders) | 2 | 4 | 2 | 3
Dystonia (Nervous system disorders) | 1 | 4 | 2 | 0
Parkinsonism (Nervous system disorders) | 3 | 1 | 5 | 1
Sedation (Nervous system disorders) | 0 | 3 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 1 | 4
Bradykinesia (Nervous system disorders) | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0
Drooling (Nervous system disorders) | 0 | 1 | 3 | 2
Dyskinesia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1 | 0 | 0
Sleep phase rhythm disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 1 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0 | 0 | 0
Head titubation (Nervous system disorders) | 0 | 1 | 0 | 0
Thermohyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0
Oculogyric crisis (Eye disorders) | 0 | 1 | 0 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 1
Auricular swelling (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 3 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1
Labile blood pressure (Vascular disorders) | 1 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3 | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0
Hunger (General disorders) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 7 | 3 | 1 | 1
Weight increased (Investigations) | 0 | 7 | 1 | 0
Blood urine present (Investigations) | 2 | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3 | 0 | 0
Blood glucose increased (Investigations) | 2 | 2 | 0 | 0
Blood cholesterol increased (Investigations) | 2 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 0
Blood pressure increased (Investigations) | 1 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 2 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 1 | 1 | 0
Low density lipoprotein increased (Investigations) | 1 | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 2
Tinea infection (Infections and infestations) | 0 | 0 | 2 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Schizophrenia (Psychiatric disorders) | 7 | 2 | 1 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 1
Thinking abnormal (Psychiatric disorders) | 0 | 0 | 0 | 1
Self-injurious ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Burnout syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 2 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1
Conjunctivitis (Eye disorders) | 1 | 1 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 9 | 9 | 13 | 8
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 4 | 3
Toothache (Gastrointestinal disorders) | 4 | 5 | 4 | 3
Abdominal discomfort (Gastrointestinal disorders) | 5 | 2 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 5 | 1
Nausea (Gastrointestinal disorders) | 8 | 6 | 4 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 3 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Dental caries (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 8 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis atrophic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lip haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 3 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1 | 2 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 3 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 1 | 1
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 3 | 1 | 4 | 1
Malaise (General disorders) | 0 | 1 | 2 | 1
Asthenia (General disorders) | 2 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 2 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 11 | 21 | 1 | 0
Irritability (General disorders) | 2 | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2 | 0
Blood prolactin increased (Investigations) | 0 | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 0 | 1
Influenza A virus test positive (Investigations) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 2
Excoriation (Injury, poisoning and procedural complications) | 4 | 1 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Chillblains (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Weight fluctuation (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 5 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nuchal rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Injection site induration (General disorders) | 4 | 6 | 0 | 0
Chest discomfort (General disorders) | 1 | 1 | 0 | 0
Injection site swelling (General disorders) | 0 | 4 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Injection site haematoma (General disorders) | 1 | 0 | 0 | 0
Injection site warmth (General disorders) | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 2 | 0 | 0
Vessel puncture site swelling (General disorders) | 1 | 0 | 0 | 0
Urobilinogen urine increased (Investigations) | 1 | 1 | 0 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood chloride increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0
Blood sodium decreased (Investigations) | 1 | 0 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1
Superficial injury of eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte percentage decreased (Investigations) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Tardive dyskinesia (Nervous system disorders) | 1 | 0 | 1 | 1
Dysstasia (Nervous system disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No